CLINICAL TRIAL: NCT04354610
Title: Prediction of Acute Heart or Kidney Injury With Cardiovascular-renal Biomarkers in Patients Hospitalised for Severe or Critical Covid-19 Infection
Brief Title: Cardiovascular and Renal Biomarkers to Predict Acute Heart or Kidney Injury in Severe Covid-19 Infection
Acronym: Nancy-CovH-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Patrick ROSSIGNOL, Prediction of Acute Heart or Kidney Injury With Cardiovascular-renal Biomarkers in Patients Hospitalised for Severe or Critical Covid-19 Infection, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020PI072
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized for Covid-19 infection (Other): Patients hospitalized for Covid-19 infection will undergo the following evaluations:
  * Clinical examination
  * Blood sample retrieved for biological assessment and biobanking
  * Telephone interview
  Interventions: Procedure: Biological samples specific to research; Procedure: Clinical examination; Procedure: Telephone follow-up

INTERVENTIONS:
Procedure: Biological samples specific to research — Blood samples, saliva collection, and urine collection to carry out biomarker assays and for the constitution of a biological collection.
Procedure: Clinical examination — Clinical examination
Procedure: Telephone follow-up — Telephone follow-up at 3 months after discharge from hospital

SUMMARY:
The Nancy Cov-H-AKI: study is a prospective, non-randomized, monocenter study performed in patients hospitalised for either the severe or the critical form of Covid-19.

The main objective of the Nancy Cov-H-AKI study is to evaluate the association of variations (from inclusion to 72H post-inclusion) of 5 blood-based cardio-vascular-renal biomarkers selected a priori, cardiac (NT-proBNP), coagulation (D-dimers), related to the renin angiotensin aldosterone system (ACE2) and renal (Penkid, and NGAL) with the appearance of acute kidney injury KDIGO grade 1 or higher OR cardiac injury in patients hospitalised for either the severe or the critical form of Covid-19

DETAILED DESCRIPTION:
Secondary objectives

Evaluate the association of the concentrations at inclusion AND of the variations (between inclusion and 72H post-inclusion) of blood and urine cardiovascular-renal biomarkers of interest (selected a priori: cardiac (NT-proBNP, (bio)-Adrenomedullin), coagulation (D-dimers), linked to the renin angiotensin aldosterone system (renin, ACE2, Angiotensin 2), inflammatory (ceramides), oxidative stress, and renal (PENKID, cystatin C) and renal glomerulo-tubulopathy ( renal functional exploration in blood and urine, and AKI (blood (NGAL, KIM-1) and urinary (IGFBP7-TIMP2)) biomarkers, AND WITHOUT a priori by an analysis of 184 blood protein biomarkers in connection with cardiovascular and inflammatory damage * ) with the appearance of:

1. AKI KDIGO grade 1 or higher or elevation of troponin >99th percentile in hospitalisation (approach with AND without a priori)
2. AKI KDIGO grade 1 or higher
3. Elevation of troponin >99th percentile in hospitalisation
4. Elevated serum creatinine >30% in hospital
5. Chronic renal failure (eDFG <60 ml / min / 1.73m2) three months after discharge from hospital
6. Cardiovascular events (stroke, myocardial infarction, hospitalization for heart failure, cardiovascular death) and mortality in hospital and at three months after discharge from hospital
7. Considering future exploratory analyses (biological collection of plasma, serum, saliva, urine, viruses) (for example other OLINK panels) on the previous endpoints

   * NGAL (Neutrophil Gelatinase Associated Lipocalin), Cystatin C, Kidney Injury Molecule-1 (Kim-1), ACE-2, renin, Brain-type Natriuretic Peptide (BNP), Adrenomedullin, FGF (fibroblast growth factor-23 are all included in the 2 Olink panels "CVDII" (https://www.olink.com/products/cvd-ii-panel/: listing) and "cardiometabolic" (https://www.olink.com/products/cardiometabolic-panel /)

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18,
* Admission for less than 3 days in the medical service (or in intensive care) for proven serious form of Covid 19 infection (respiratory rate >30 / min, or desaturation in air ≤ 93%, or PaO2 / FiO2 ≤ 300mmHg)
* OR Admission for less than 2 days in intensive care (or resuscitation intensive care) for critical form of Covid 19 (shock or respiratory failure).
* GFR greater than 30 ml / min / 1.73m2.
* Troponin <99th percentile.
* Patient affiliated to a social security scheme or beneficiary of such a scheme
* The patient or their representative received complete information on the study and signed and dated the emergency situation informed consent/inclusion form in accordance with article L1122-1-3 of the French Public Health Code (Code de la Santé Publique).

Exclusion Criteria:

Exclusion criterion for patients taking part in clinical research.

* AKI KDIGO grade 1 on the day of visit 1
* Pregnant women, parturient, or nursing mothers
* A person of full age subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person deprived of their liberty by a judicial or administrative decision,
* Person undergoing psychiatric treatment under articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Worsening of renal function by at least KDIGO grade 1 during hospitalization for Covid-19 infection | From inclusion to hospital discharge, an average of 21 days
  Composite endpoint : Worsening of renal function by at least KDIGO grade 1 criteria from inclusion visit OR troponin greater than 99th percentile during hospitalization for Covid-19 infection (with Outcome 2).
Troponin greater than 99th percentile during hospitalization for Covid-19 infection | From inclusion to hospital discharge, an average of 21 days
  Composite endpoint : Worsening of renal function by at least KDIGO grade 1 criteria from inclusion visit OR troponin greater than 99th percentile during hospitalization for Covid-19 infection (with Outcome 1)

SECONDARY OUTCOMES:
AKI KDIGO grade 1 or higher in hospitalisation (approach with AND without a priori) | From inclusion to hospital discharge, an average of 21 days
  Composite endpoint : AKI KDIGO grade 1 or higher or Elevation of troponin> 99th percentile in hospitalisation (approach with AND without a priori) ((with Outcome 3 )
Elevation of troponin> 99th percentile in hospitalisation (approach with AND without a priori) | From inclusion to hospital discharge, an average of 21 days
  Composite endpoint : AKI KDIGO grade 1 or higher or Elevation of troponin> 99th percentile in hospitalisation (approach with AND without a priori) (with Outcome 3)
AKI KDIGO grade 1 or higher | From inclusion to hospital discharge, an average of 21 days
  AKI KDIGO grade 1 in hospitalisation
Association with troponin elevation >99th | From inclusion to hospital discharge, an average of 21 days
  Association with troponin elevation >99th percentile during hospitalisation
Association with elevation of serum creatinine >30% | From inclusion to hospital discharge, an average of 21 days
  Association with elevation of serum creatinine >30% during hospitalisation
With the onset of chronic renal failure (eDFG <60 ml / min / 1.73m2) | 3 months after discharge from hospital
  With the onset of chronic renal failure (eDFG <60 ml / min / 1.73m2) three months after discharge from hospital
The occurrence of cardiovascular events (stroke, myocardial infarction, hospitalisation for heart failure, cardiovascular death) during hospitalisation and three months after discharge from hospital | From inclusion to three months after discharge from hospital
  Composite outcome : the occurrence of cardiovascular events (stroke, myocardial infarction, hospitalisation for heart failure, cardiovascular death) and death from any cause during hospitalisation and three months after discharge from hospital
The occurrence of death from any cause during hospitalisation and three months after discharge from hospital | From inclusion to three months after discharge from hospital
  Composite outcome : the occurrence of cardiovascular events (stroke, myocardial infarction, hospitalisation for heart failure, cardiovascular death) and death from any cause during hospitalisation and three months after discharge from hospital

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Nancy, Nancy
  - CHRU de Nancy, Vandœuvre-lès-Nancy